CLINICAL TRIAL: NCT00059033
Title: Clinical Laboratory Evaluation of Primary Chronic Autonomic Failure
Brief Title: Evaluation of Primary Chronic Autonomic Failure
Status: Terminated | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030004; 03-N-0004
Record Dates: First submitted 2003-04-16; First posted 2003-04-16 (Estimated); Last update posted 2019-12-12 (Actual); Status verified 2018-10-30

CONDITIONS: Autonomic Nervous System Diseases
Keywords: 6-[18F]Fluorodopamine; Autonomic Failure; Parkinson's Disease; Multiple System Atrophy; Pure Autonomic Failure; Primary Chronic Autonomic Failure; CAF
MeSH Terms: conditions — Autonomic Nervous System Diseases; Pure Autonomic Failure; Parkinson Disease; Multiple System Atrophy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No

SUMMARY:
This study will conduct tests in patients with primary chronic autonomic failure (CAF) to learn more about these disorders, which include pure autonomic failure, multiple system atrophy, Parkinson's disease with autonomic failure, and autoimmune autonomic neuropathy.

Healthy volunteers and patients with primary CAF 18 years of age or older may be eligible for this study. Participants undergo some of the following tests:

* Blood studies, including arterial catheter insertion to measure blood pressure and collect arterial blood samples, blood flow studies using sensors applied to the skin and a pressure cuff around a limb, and blood draw for genetic studies.
* Bladder motility: Ultrasound test of bladder function.
* Electrocardiogram and heart ultrasound.
* Responses to changes in temperature: Warm water and then room temperature water are passed through watertight pads applied to the back and front of the body and body temperatures are measured.
* Gastrointestinal motility: Bowel sounds are recorded using a microphone placed on the abdomen.
* Lower body negative pressure: The lower body is placed into an airtight barrel-like chamber. Some air is sucked out of the barrel, causing blood to pool in the legs, as occurs during standing.
* Lumbar puncture: A needle is inserted in the space between the bones in the lower back to collect a small sample of cerebrospinal fluid.
* Microdialysis to measures levels of chemicals in the body fluid of certain tissues. A solution is passed through a thin tube inserted into the skin. Chemicals in the body tissues enter the solution. The solution is collected and the chemical levels are measured.
* PET scanning: A nuclear medicine test to produce images of body organs. For patients with urinary problems, a catheter is inserted into the bladder before starting the scan.
* Pupillometry: The pupil of the eye is measured using a special camera in a light-controlled room.
* QSART. A small amount of a brain chemical is applied to the skin with a tiny amount of electricity, and the sweat in a nearby patch of skin is measured.
* Measurement of saliva production, using a cotton-like material placed between the teeth and gums to absorb saliva.
* Skin electrical conduction test, using sensors on the skin to measure sweat production.
* Skin and core temperature measurements using sensors on the skin and in the ear canal.
* Speech and swallowing assessment for patients with speech and swallowing difficulties.
* Stress echocardiogram: A catheter is placed in the subject's arm for sampling blood or giving a drug while the subject exercises. During the test, blood pressure, pulse rate, and EKG are continuously monitored.

DETAILED DESCRIPTION:
Objective:

In dysautonomias, altered functions of one or more components of the autonomic nervous system adversely affect health. Primary dysautonomias have been classified clinically into chronic autonomic failure (CAF) syndromes that include pure autonomic failure (PAF), multiple system atrophy (MSA), and Parkinson disease (PD) with autonomic failure (manifested especially by neurogenic orthostatic hypotension (OH)). Clinical assessment alone is often inadequate for correct diagnosis and does not provide insights into mechanisms or identify new therapeutic targets. This protocol calls for continuous development and assessment of physiological, neuropharmacologic, neurochemical, neuroimaging, and other clinical laboratory approaches, to identify lesion types and sites in CAF and improve diagnosis, increase mechanistic understanding, and incite novel therapeutics. PAF, MSA, and PD exemplify alpha synucleinopathies, in which deposits of the protein alpha-synuclein occur in Lewy bodies in catecholamine-producing neurons (PD, PAF) or in the cytoplasm of glial cells (MSA). Only the Lewy body forms of synucleinopathy are consistently associated with loss of catecholaminergic neurons. Under this protocol we have obtained evidence that patients with Lewy body diseases have decreased ability to take up intra-neuronal catecholamines from the cytoplasm into storage vesicles. Cytoplasmic catecholamines are cytotoxic, such as by enzyme-catalyzed conversion to highly reactive catecholaldehydes. By studying CAF patients we hope to make discoveries that will yield a unifying, integrative concept for the pathogenesis and different clinical manifestations of Lewy body diseases. Autonomic function testing under this protocol is also required for screening purposes for entry into other protocols of the Clinical Neurocardiology Section. Moreover, comprehensive autonomic function testing is requested in patients of the NIH Undiagnosed Diseases Program. Finally, in a long-term project as a member of the Autonomic Rare Diseases Clinical Research Consortium we are applying this testing to study the natural history of neurogenic OH.

Study Population:

The study population consists of patients with idiopathic, or primary, CAF, with emphasis on PAF, MSA, and PD. Comparison groups include healthy volunteers (HVs), patients with PD who do not have OH, and patients with iatrogenic CAF such as from bilateral thoracic sympathectomies.

Design: Subjects undergo multiple physiological, neuropharmacologic, neurochemical, and neuroimaging, and other tests, to see if the results by different modalities agree and point to specific sites and types of lesions.

Outcome Measures:

Physiological outcome measures include hemodynamic responses to the Valsalva maneuver, orthostasis, and altered temperature at skin of the back. Neuropharmacologic measures include cardiovascular responses to test drugs that probe specific components of the autonomic nervous system. Neurochemical measures include plasma, cerebrospinal fluid, microdialysate, urine, and skin biopsy tissue levels of catecholamines and related compounds. Neuroimaging measures include positron emission tomographic scanning after injection of 18F-dopamine, 18F-DOPA, 13N-ammonia, or 11C-methylreboxetine.

ELIGIBILITY:
* INCLUSION CRITERIA:

The subjects are patients with known or suspected primary CAF, based on referral information and confirmation of the clinical diagnosis at the intake evaluation. They are classified by results of the intake evaluation and then undergo comprehensive autonomic function testing.

Patients with primary or iatrogenic CAF are included. Control patients have been previously diagnosed with PD or MSA without OH, confirmed at the time of the intake evaluation.

Healthy Volunteers 18 years old or older are included. People at increased risk for PD or CAF consent in this study as if they were patients (e.g., to enable DNA extraction and storage).

All subjects must be able to provide their own consent to participate or have an existing Durable Power of Attorney (DPA) in place.

EXCLUSION CRITERIA:

Age: People younger than 18 years old are excluded.

Risk: A candidate subject is excluded if, in the judgment of the Principal Investigator or Clinical Director, protocol participation would place the subject at substantially increased acute medical risk. This includes the risks associated with air travel to the NIH. A candidate subject is excluded if, in the opinion of the Principal Investigator or Clinical Director, the medical risk outweighs the potential scientific benefit.

Disqualifying Conditions A candidate subject is excluded if there is a disqualifying condition. Examples of disqualifying conditions are hepatic or renal failure (defined by serum creatinine more than 1.5 g/dL), symptomatic congestive heart failure, severe anemia, psychosis, refractory ventricular arrhythmias, and symptomatic coronary heart disease. Patients are excluded from further participation if the results of the intake evaluation lead to a diagnosis of a secondary form of CAF, such diabetic autonomic neuropathy. Candidate subjects who are unable to give their own consent and who do not have an existing DPA in place are excluded. Pregnant or lactating women are excluded from the study.

Medications Patients with known or suspected allergy or hypersensitivity to any test drug are excluded from receiving that drug. Patients are not to discontinue any medications before the patient or the patient s doctor discusses this with the Principal Investigator, Research Nurse, or Nurse Practitioner. If it is decided that discontinuing medications would be unsafe, then the patient may be excluded from all or part of the study.

Herbal Medicines and Dietary Supplements Certain herbal medicines or dietary supplements are known or suspected to interfere with the experimental results, and such herbal medicines or dietary supplements may be disallowed before enrollment in the study. For many herbal medicines or dietary supplements, the mechanisms of action and therefore the possible effects on the experimental results are unknown. In cases where the subjects wish to continue their herbal medicines or dietary supplements while on study, and search of the available medical literature fails to identify effects that are known or expected to interfere with the experimental results, then the subjects may participate.

Practical Limitations Patients in whom we feel it would be difficult to insert a catheter into a vein may be excluded. Subjects who are not expected clinically to tolerate lying still during the procedures may be excluded.

Pregnancy Pregnant or lactating women are excluded from the protocol overall. In women with child-bearing potential, blood testing for pregnancy will be done with 24 hours before initial testing (except for obtaining the medical history and physical examination) or any testing involving radioactivity under the protocol. Repeat pregnancy testing will be done before any procedure or drug administration under the protocol that takes place more than one week from a previous pregnancy test. Participants will not start or remain in the study if pregnancy test is positive.

Refusal to Undergo Certain Procedures Candidate subjects are excluded if they refuse to undergo certain procedures. These are: (1) IV catheter; (2) electrocardiogram; (3) blood drawing; (4) DNA extraction and storage (patients and non-HV controls only); and (5) DNA analysis (patients and non-HV controls only).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 325 (Actual)
Dates: Start 2003-04-10; Study Completion 2018-10-30

CONTACTS AND LOCATIONS:
Overall Officials: David S Goldstein, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Gilman S, Low P, Quinn N, Albanese A, Ben-Shlomo Y, Fowler C, Kaufmann H, Klockgether T, Lang A, Lantos P, Litvan I, Mathias C, Oliver E, Robertson D, Schatz I, Wenning G. Consensus statement on the diagnosis of multiple system atrophy. American Autonomic Society and American Academy of Neurology. Clin Auton Res. 1998 Dec;8(6):359-62. doi: 10.1007/BF02309628. PMID 9869555
- [Background] Low PA, Gilden JL, Freeman R, Sheng KN, McElligott MA. Efficacy of midodrine vs placebo in neurogenic orthostatic hypotension. A randomized, double-blind multicenter study. Midodrine Study Group. JAMA. 1997 Apr 2;277(13):1046-51. PMID 9091692
- [Background] Reinhardt MJ, Jungling FD, Krause TM, Braune S. Scintigraphic differentiation between two forms of primary dysautonomia early after onset of autonomic dysfunction: value of cardiac and pulmonary iodine-123 MIBG uptake. Eur J Nucl Med. 2000 May;27(5):595-600. doi: 10.1007/s002590050548. PMID 10853817